CLINICAL TRIAL: NCT05631080
Title: Anatomical Endoscopic Enucleation of the Prostate for Treatment of Bladder Outlet Obstruction in Patients With Low-risk Prostate Cancer on Surveillance Protocol, Prospective Assessment of Functional and Oncological Outcome
Brief Title: Transurethral Prostate Enucleation in Surveillance Protocol for Low Risk Prostate Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed Elshal, A. Professor of Urology, Mansoura University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mans 22-4-2016
Record Dates: First submitted 2022-11-19; First posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Prostate Cancer Stage I; Bladder Outlet Obstruction
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Bladder Neck Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surveillance with medical treatment for bladder outlet obstruction (No Intervention): Patients with low-risk prostate cancer who were elected for active surveillance protocol will have only medical treatment for control of their lower urinary tract symptoms secondary to bladder outlet obstruction
- Surveillance with anatomical endoscopic enucleation of the prostate for bladder outlet obstruction (Active Comparator): Patients with low-risk prostate cancer who were elected for active surveillance protocol will be offered anatomical endoscopic enucleation of the prostate for control of their lower urinary tract symptoms secondary to bladder outlet obstruction
  Interventions: Procedure: Anatomical Endoscpic enucleation of the Prostate

INTERVENTIONS:
Procedure: Anatomical Endoscpic enucleation of the Prostate — Transurethral endoscopic enucleation of the prostate adenoma
  Other Names: AEEP
  Arms: Surveillance with anatomical endoscopic enucleation of the prostate for bladder outlet obstruction

SUMMARY:
We will compare oncological and functional outcomes of anatomical endoscopic enucleation of the prostate (AEEP) versus continued medical treatment in low-risk prostate cancer patients for whom an active surveillance protocol was selected.

DETAILED DESCRIPTION:
Prostate cancer is the most common cancer in men; in 2018 1,276,106 new cases of prostate cancer were reported worldwide (1).

The diagnosis of prostate cancer is based on the microscopic evaluation of prostate tissue obtained via needle biopsy.

The International Society of Urological Pathology (ISUP) Consensus system assigns new Grade Groups from 1 to 5, derived from the Gleason score (2).

Clinicians have stratified the diagnosis into low, intermediate, and high-risk disease based on the sum of Gleason patterns, prostate specific antigen (PSA) level, and clinical stage (3).

Recently The National Comprehensive Cancer Network risk stratification uses a 5-tier system by adding very low- and very high- as a subdivision of the low- and high-risk groups (4).

Men diagnosed with localized disease (defined as no regional lymph nodes or distant metastases) have 3 primary options: expectant management, surgery and radiation.

Expectant management (monitoring for prostate cancer progression while not undergoing definitive therapy) consists of watchful waiting and active surveillance (5).

According to The Prostate Testing for Cancer and Treatment (ProtecT) trial which randomized 1643 localized prostate cancer men to active monitoring, surgery, or radiation. At 120 months, ProtecT found that 1.5% of patients on active monitoring died from prostate cancer, which did not differ significantly from the 0.9% after surgery or the 0.7% after radiation (6).

The use of active surveillance (AS) for men with low-risk prostate cancer (PCa) is well established, although the criteria for admission to a protocol vary according to the institution. (7-9) Men with significantly enlarged prostates (>100 g) may be assigned a high-risk category when their prostate-specific antigen (PSA) rises above 10 ng/ml, although there is evidence AS is safe in this population. (10) In the presence of lower urinary tract symptoms (LUTS), men with significantly enlarged prostates often undergo radical prostatectomy (RP) to treat PCa and coexisting LUTS. This approach, which prioritizes oncologic control, may increase surgical morbidity for patients who otherwise might continue AS after an outlet procedure to address their LUTS.

The use of holmium laser enucleation of the prostate (HoLEP) for the management of LUTS in men with significantly enlarged prostates and coexisting low-risk PCa has not been prospectively studied. HoLEP has proven to be a safe and effective treatment for men with LUTS. (11) Incidental detection of malignancy at the time of HoLEP ranges from 5% to 13% in men without a prior diagnosis of PCa, and there is evidence PSA has improved sensitivity for cancer progression in the post-HoLEP setting. (12-15) The management of T1a-b PCa incidentally discovered after transurethral resection of prostate (TURP) has been well documented with AS recommended for most patients. (16-18) However, the management of men with known low-risk PCa, clinically significant LUTS, and significantly enlarged prostates remains underexplored.

Herein, we prospectively assess patients with low-risk PCa on AS who underwent AEEP for clinically significant LUTS and enlarged prostate gland size.

Our study focuses on functional and oncologic outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Life expectancy >/= 10 years
2. Low risk prostate cancer with minor institutional amendment of EAU guidelines:

   * PSA < 10 ng/ml or up to 20 ng/ml if PSA density is more than 15%
   * Stage T1, T2a.
   * Gleason score <7 (ISUP grade 1)
3. Bladder outlet obstruction:

   * IPSS > 9
   * Peak flow rate (Qmax < 15)
   * Imperative indication for BOO surgery

Exclusion criteria:

* Patients who are not willing
* Patients with bladder dysfunction (cystopathy) or other infravesical cause of obstruction other than prostate

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — prostate disorder only in males
Enrollment: 50 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2022-09 (Actual); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
PSA progression | one year
  changes of PSA level from baseline to one year follow up following active treatment
radiological progression | one year
  cancer progression as depicted by multiparametric MRI

SECONDARY OUTCOMES:
relief of bladder outlet obstruction | one year
  improvement of urine flow parameters as depicted by peak flow rate (ml/sec)
relief of lower urinary tract symptoms | one year
  improvement of urinary symptoms as depicted by symptom score (International prostate symptom score)
2 years progression free survival | 2 years
  PSA, Radiological and grade progression whenever biopsy is indicated
5 years progression free survival | 5 years
  PSA, Radiological and grade progression whenever biopsy is indicated

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elshal, MD, Principal Investigator — Mansoura University
Locations (1):
- Urology and nephrology center, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: No